CLINICAL TRIAL: NCT07183930
Title: Comparison Between Tubeless and Tube Percutaneous Nephrolithotomy in Pediatric Population: A Randomized Controlled Trial
Brief Title: Tubeless vs Tube PCNL in Pediatric Nephrolithiasis: A Randomized Controlled Trial.
Acronym: TUBELESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr. Waseem Ullah, Tariq, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMC-IREB-533
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Nephrolithiasis; Kidney Stones; Pediatric Nephrolithiasis
Keywords: Blood transfusion; Kidney stone surgery; Tubeless PCNL; PCNL; Percutaneous nephrolithotomy; Stone-free rate
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubeless PCNL (Experimental): Percutaneous nephrolithotomy (PCNL) performed without nephrostomy tube placement. After complete stone clearance and confirmation of hemostasis, only a double-J stent is placed; the access tract is left to seal naturally.
  Interventions: Procedure: Tubeless Percutaneous Nephrolithotomy (PCNL)
- Tube PCNL (Active Comparator): Standard PCNL performed with placement of a nephrostomy tube following stone clearance, along with a double-J stent.
  Interventions: Procedure: Standard Tube Percutaneous Nephrolithotomy (PCNL)

INTERVENTIONS:
Procedure: Tubeless Percutaneous Nephrolithotomy (PCNL) — Mini-PCNL with tract dilation up to 18 Fr and stone fragmentation by pneumatic lithotripsy. Following clearance, a double-J stent is placed; no nephrostomy tube is inserted.
  Arms: Tubeless PCNL
Procedure: Standard Tube Percutaneous Nephrolithotomy (PCNL) — Mini-PCNL with tract dilation up to 18 Fr and stone fragmentation by pneumatic lithotripsy. Following clearance, a 14 Fr nephrostomy tube and a double-J stent are placed.
  Arms: Tube PCNL

SUMMARY:
This study is designed to compare two surgical techniques for removing kidney stones in children and adolescents (ages 6-18 years). Both methods are types of percutaneous nephrolithotomy (PCNL), a standard procedure for kidney stones larger than 10 mm.

In the traditional method, a temporary tube (nephrostomy tube) is left in the kidney after surgery to drain urine. In the newer "tubeless" method, the tube is not used, and only a small internal stent may be placed. We want to find out if the tubeless method is as safe and effective as the traditional method, and whether it reduces pain, hospital stay, and the need for blood transfusions. The study involves 640 patients at Khyber Teaching Hospital in Peshawar, Pakistan. Each participant is randomly assigned to one of the two techniques.

DETAILED DESCRIPTION:
Pediatric kidney stones are increasingly common and often require surgical management when stones are larger than 10 mm or fail to pass with conservative treatment. Percutaneous nephrolithotomy (PCNL) is the gold standard for such cases. Traditionally, PCNL involves the placement of a nephrostomy tube to ensure postoperative drainage. However, this tube can increase discomfort, lengthen hospital stay, and sometimes lead to bleeding.

Recent advances in adult populations suggest that "tubeless" PCNL-where no external drainage tube is left-may reduce postoperative pain, decrease hospital stay, and improve recovery, without compromising safety. Evidence in children remains limited, mostly from small retrospective series.

This randomized controlled trial was conducted at Khyber Teaching Hospital, Peshawar, between October 2024 and March 2025. A total of 640 pediatric patients aged 6-18 years with renal stones >10 mm were randomized into two groups: Group A (Tubeless PCNL, n=320) and Group B (Tube PCNL, n=320). All procedures were performed by a single experienced pediatric urologist using standardized mini-PCNL techniques.

The primary outcomes include operative time, hospital stay, blood transfusion requirement, and stone-free status on discharge. Secondary outcomes include postoperative pain scores, analgesic use, complications (graded by Clavien-Dindo classification), time to resumption of normal activities, and patient/family satisfaction.

By directly comparing the two approaches in a large pediatric cohort, this study provides high-quality evidence to determine whether tubeless PCNL should be considered the preferred technique in appropriately selected children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 18 years
* Either gender
* Renal calculi larger than 10 mm on imaging
* Failed conservative management or extracorporeal shock wave lithotripsy (ESWL)
* Normal renal function
* Informed consent from parents/guardians
* Assent from children aged 12 years and above

Exclusion Criteria:

* Prior renal surgery or ureteral stenting
* Congenital urological anomalies
* Active urinary tract infection at the time of surgery
* Known bleeding disorders or use of anticoagulant medication
* Significant comorbid medical conditions
* Pregnancy (in adolescent females)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 640 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay (days) | From surgery to discharge (up to 7 days).
  Number of days from the date of surgery until discharge from hospital.
Operative time (minutes) | During surgery (single procedure).
  Duration of the surgical procedure measured from skin incision to skin closure, recorded in minutes.
Blood transfusion requirement (%) | surgery through hospital discharge (up to 7 days).
  Proportion of participants requiring perioperative blood transfusion, as documented in patient records.
Stone-free status (%) | At hospital discharge (within 48 hours after surgery).
  Proportion of patients with no residual stone fragments >2 mm on postoperative imaging (ultrasound or CT).

SECONDARY OUTCOMES:
Postoperative pain score (VAS) | First 24 hours post-surgery
  Pain intensity assessed using the Visual Analog Scale (0-10), averaged over the first 24 hours after surgery.
Analgesic requirement (morphine equivalents, mg) | First 48 hours post-surgery
  Total opioid dose used postoperatively in the first 48 hours, converted to morphine equivalents and measured in milligrams.
Postoperative complications (Clavien-Dindo classification) | surgery to discharge (up to 7 days)
  Number and severity of complications graded using the Clavien-Dindo classification system.
Time to return to normal activity (days) | Up to 30 days post-surgery
  Number of days from surgery until the patient resumes routine daily activities, as reported by patient/parent.
Patient and family satisfaction score | At hospital discharge (within 7 days post-surgery)
  Satisfaction with overall care and outcome, measured using a 10-point Likert scale questionnaire completed at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ahmad, MBBS, FCPS, Principal Investigator — Khyber Teaching Hospital, Peshawar
Locations (1):
- Khyber Teaching Hospital, Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing plans have not been finalized. This will depend on journal requirements, funding agency policies, and institutional guidelines at the time of publication.